CLINICAL TRIAL: NCT05879497
Title: 68Ga-NY104 PET/CT in Patients With Metastasis/Recurrence Clear Cell Renal Cell Carcinoma Suspicion: a Prospective, Single Center, Single Arm Imaging Trial
Brief Title: 68Ga-NY104 PET/CT in Patients With Metastasis/Recurrence Clear Cell Renal Cell Carcinoma Suspicion
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NYCRMS
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: 68Ga-NY104; PET/CT; Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-NY104 PET/CT (Experimental): Each patient will receive one dose of 68Ga-NY104 by intravenous route. Dedicated whole-body PET/CT imaging will be performed.
  Interventions: Diagnostic Test: 68Ga-NY104 PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-NY104 PET/CT — Participants will be administered a single, intravenous bolus of 68Ga-NY104 The recommended administered activity of 68Ga-NY104 is 1.8-2.2 MBq per kilogram bodyweight, subject to variation that may be required owing to variable elution efficiencies obtained during the lifetime of the 68Ga / 68Ga generator The CT and PET imaging session will begin approximately 45 to 75 minutes after 68Ga-NY104 administration.
  Other Names: 68Ga-NYM005 PET/CT

SUMMARY:
This is a prospective, single-center, single-arm phase 2 study in patients with clear cell renal cell carcinoma and metastasis or recurrence suspicion. The goal is to determine the sensitivity and specificity of 68Ga-NY104 PET/CT in patients with clear cell renal cell carcinoma and metastasis or recurrence suspicion

DETAILED DESCRIPTION:
This is a prospective, single-center, single-arm phase 2 study in patients with clear cell renal cell carcinoma and metastasis or recurrence suspicion. Each patient will receive one dose of 68Ga-NY104. Dedicated whole-body PET/CT imaging will be performed. PET/CT studies will be interpreted by two readers, both of whom will provide independent and blinded interpretations. Imaging interpretations and a composite ground truth will be used to estimate the diagnostic efficacy of 68Ga-NY104 PET/CT.

A total of 40 patients will be recruited at Peking Union Medical College Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 y
2. Histopathological diagnosis of clear cell renal cell carcinoma
3. Suspected of metastasis or recurrence from ccRCC based on previous conventional imaging or 18F-FDG PET/CT scan.
4. Expected survival of at least 6 months
5. ECOG ≤ 2
6. Written informed consent provided for participation in the trial
7. In the opinion of investigator, willing and able to comply with required study procedures.

Exclusion Criteria:

1. On VEGF TKI treatment less than 1 week before 68Ga-NY104 PET/CT. TKI is known to affect girentuximab binding in patients with ccRCC and is expected to have the same effect on 68Ga-NY104. If patients were on VEGF TKI treatment, such as sunitinib, sorafenib, cabozantinib, pazopanib, or lenvatinib, a washout of one week before 68Ga-NY104 PET/CT is required.
2. Patients on HIF antagonist treatment < 3 months before 68Ga-NY104 PET/CT. CA9, which encodes carbonic anhydrase IX (CAIX), is one of the genes most strongly upregulated by HIF-1. HIF antagonist, such as Belzutifan, might affect the expression of CAIX and thus the binding of 68Ga-NY104 to tumor. Withdraw of at least 3 months is required for HIF antagonist.
3. Pregnancy or breastfeeding.
4. Severe claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Binary reading of lesions identified on 68Ga-NY104 PET/CT | From study completion to 1 month after completion
  Any focal accumulation in the lesion suspected of metastasis or recurrence that cannot be explained by physiologic uptake of 68Ga-NY104 will be interpreted as PET positive.

CONTACTS AND LOCATIONS:
Overall Officials: Li Huo, MD, Principal Investigator — Peking Uion Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Available upon request
Supporting Information: Study Protocol
Time Frame: Within 2 years after the publication of the main results
Access Criteria: No limit.